CLINICAL TRIAL: NCT04507724
Title: The Use of Biochemical Analyzes to Monitor the Development of Wounds: Part 1: Analysis of Wounds Without VAC Therapy: Part 2: Analysis of Wound Fluids Under VAC Therapy
Brief Title: The Use of Biochemical Analyzes to Monitor the Development of Wounds
Acronym: NPWW
Status: Completed | Type: Observational
Sponsor: Qualizyme Diagnostics GmbH & Co KG (Industry)
Responsible Party: Principal Investigator, Christina Helene Wolfsberger, Sub-Investigator, Medical University of Graz
Other Study IDs: NPWW
Record Dates: First submitted 2020-07-22; First posted 2020-08-11 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Wound; Wound Infection; Wound Contamination; Diagnostic Techniques and Procedures; Negative Pressure Wound Therapy; Biomarker
Keywords: wound infection; negative pressure wound therapy; diagnostic tool; biomarker
MeSH Terms: conditions — Wounds and Injuries; Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic wounds represent a growing challenge in medical care.

Part 1: The aim of this part of the study was to collect wound swabs and to answer the question whether the rapid diagnostic tool using enzyme activities can display an infection prematurely. This means that an increased enzyme activity (especially MPO, NHE, LYS, gelatinase, pH) measured overed 3 days, would indicate a change in the wound bed (infection, Inflammation) earlier than the regularly performed clinical assessment.

Part 2: The aim of this part of the study was to evaluate (I) the possibility of wound fluid acquisition by means of an "additional collector" during ongoing NPWT and to answer if (II) this secretion can be biochemically analyzed for enzyme activities in order to be able to detect a change in the wound situation at an early stage.

DETAILED DESCRIPTION:
The study is composed of two parts, which run independently of each other. However, in both parts the course of the wounds is analyzed.

Part 1: Two wound swabs are taken. One used for routinely performed microbiological analysis and the second will be used for biochemical analysis (enzyme activities). The aim of the wound swabs is to answer the question whether the rapid diagnostic tool used in the examination can display an infection prematurely or not. This means that an increased enzyme activity (especially MPO, NHE, LYS, gelatinase, pH) would indicate a change in the wound bed (infection, inflammation) earlier than the regular clinical assessment. These wound swabs are expected to function as an improvement of the biochemical assays or rather of the technology concerning sensitivity and specificity of, for example, the pH number, the MPO, the LYS, the gelatinase and the elastase. In addition to that, the correlation between the Enzyme activities and the course of the infection will be examined. This technology is supposed to be later used as an early infection diagnostic tool in wound fluids. The followup of this testing system is a crucial prerequisite for the application of the technology in VAC therapy (part 2).

Part 2: The findings of this examination will be used to investigate the applicability of the developed in-vitro early infection diagnostic tool in negative-pressure therapy (VAC therapy; vacuum assisted closure).

Patients of the plastic surgery with a NPWT are included in this prospective study. Before the NPWT will be applied, two swabs (biochemical and microbiological analysis) of the wounds will be taken. After installation of the dressing, the connecting tube between the wound and the vacuum-generating device will be cut and an "additional collector" will be inserted. This collector will be changed daily and afterwards the concentrations of enzymes (lysozyme, elastase, myeloperoxidase) will be biochemically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* older than 18 years old
* open wound of varying etiology
* VAC therapy (KCI) (part 2)

Exclusion Criteria:

* under 18 years old
* pregnant women
* less than three measurement data (less than three swabs) = part 1
* VAC-instill therapy = part 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected by inpatients with wounds (part 1) or with negative pressure wound therapy (part 2)
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Part 1: biochemical analysis of wounds | during hospitalization
  Elevated enzyme activities (biochemical analysis of wound swabs) give information of the condition of the wound bed (infection, inflammation).
Part 2: Descriptive assessment of the feasibility of collecting wound fluid during ongoing negative pressure wound therapy | during negative pressure wound therapy
  The aim is to answer the question if it is feasible to collect wound fluid during ongoing negative pressure wound therapy and analyze this wound fluid biochemically.

SECONDARY OUTCOMES:
Part 2: Evaluating changes in enzyme activities in the collected wound fluid | Starting immediately after installation of the negative-pressure dressing and lasting for 3 days.
  The collected wound fluid will be analyzed biochemically daily over three days. This might give as informations of wounds as an "in-vitro early infection diagnostic tool"

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schintler, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Division of Plastic, Aesthetic and Reconstructive Surgery, Department of Surgery, Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] McDaniel JC, Roy S, Wilgus TA. Neutrophil activity in chronic venous leg ulcers--a target for therapy? Wound Repair Regen. 2013 May-Jun;21(3):339-51. doi: 10.1111/wrr.12036. Epub 2013 Mar 28. PMID 23551462
- [Background] Trengove NJ, Bielefeldt-Ohmann H, Stacey MC. Mitogenic activity and cytokine levels in non-healing and healing chronic leg ulcers. Wound Repair Regen. 2000 Jan-Feb;8(1):13-25. doi: 10.1046/j.1524-475x.2000.00013.x. PMID 10760211
- [Background] Ladwig GP, Robson MC, Liu R, Kuhn MA, Muir DF, Schultz GS. Ratios of activated matrix metalloproteinase-9 to tissue inhibitor of matrix metalloproteinase-1 in wound fluids are inversely correlated with healing of pressure ulcers. Wound Repair Regen. 2002 Jan-Feb;10(1):26-37. doi: 10.1046/j.1524-475x.2002.10903.x. PMID 11983004
- [Background] Yager DR, Zhang LY, Liang HX, Diegelmann RF, Cohen IK. Wound fluids from human pressure ulcers contain elevated matrix metalloproteinase levels and activity compared to surgical wound fluids. J Invest Dermatol. 1996 Nov;107(5):743-8. doi: 10.1111/1523-1747.ep12365637. PMID 8875960
- [Background] Izadi K, Ganchi P. Chronic wounds. Clin Plast Surg. 2005 Apr;32(2):209-22. doi: 10.1016/j.cps.2004.11.011. PMID 15814118
- [Background] Argenta LC, Morykwas MJ. Vacuum-assisted closure: a new method for wound control and treatment: clinical experience. Ann Plast Surg. 1997 Jun;38(6):563-76; discussion 577. PMID 9188971
- [Background] James GA, Swogger E, Wolcott R, Pulcini Ed, Secor P, Sestrich J, Costerton JW, Stewart PS. Biofilms in chronic wounds. Wound Repair Regen. 2008 Jan-Feb;16(1):37-44. doi: 10.1111/j.1524-475X.2007.00321.x. Epub 2007 Dec 13. PMID 18086294
- [Background] Steenvoorde P, van Engeland A, Oskam J. Vacuum-assisted closure therapy and oral anticoagulation therapy. Plast Reconstr Surg. 2004 Jun;113(7):2220-1. doi: 10.1097/01.prs.0000123603.32963.11. No abstract available. PMID 15253223
- [Background] Morykwas MJ, Argenta LC, Shelton-Brown EI, McGuirt W. Vacuum-assisted closure: a new method for wound control and treatment: animal studies and basic foundation. Ann Plast Surg. 1997 Jun;38(6):553-62. doi: 10.1097/00000637-199706000-00001. PMID 9188970
- [Background] Huang C, Leavitt T, Bayer LR, Orgill DP. Effect of negative pressure wound therapy on wound healing. Curr Probl Surg. 2014 Jul;51(7):301-31. doi: 10.1067/j.cpsurg.2014.04.001. Epub 2014 Apr 26. PMID 24935079
- [Background] Nuutila K, Yang L, Broomhead M, Proppe K, Eriksson E. Novel negative pressure wound therapy device without foam or gauze is effective at -50 mmHg. Wound Repair Regen. 2019 Mar;27(2):162-169. doi: 10.1111/wrr.3. Epub 2018 Oct 31. PMID 30378215
- [Background] Isago T, Nozaki M, Kikuchi Y, Honda T, Nakazawa H. Effects of different negative pressures on reduction of wounds in negative pressure dressings. J Dermatol. 2003 Aug;30(8):596-601. doi: 10.1111/j.1346-8138.2003.tb00441.x. PMID 12928528
- [Background] Fleischmann W, Russ M, Westhauser A, Stampehl M. [Vacuum sealing as carrier system for controlled local drug administration in wound infection]. Unfallchirurg. 1998 Aug;101(8):649-54. doi: 10.1007/s001130050318. German. PMID 9782769
- [Background] Timmers MS, Graafland N, Bernards AT, Nelissen RG, van Dissel JT, Jukema GN. Negative pressure wound treatment with polyvinyl alcohol foam and polyhexanide antiseptic solution instillation in posttraumatic osteomyelitis. Wound Repair Regen. 2009 Mar-Apr;17(2):278-86. doi: 10.1111/j.1524-475X.2009.00458.x. PMID 19320897
- [Background] Blokhuis-Arkes MH, Haalboom M, van der Palen J, Heinzle A, Sigl E, Guebitz G, Beuk R. Rapid enzyme analysis as a diagnostic tool for wound infection: Comparison between clinical judgment, microbiological analysis, and enzyme analysis. Wound Repair Regen. 2015 May-Jun;23(3):345-52. doi: 10.1111/wrr.12282. Epub 2015 Jun 19. PMID 25816836
- [Background] Hasmann A, Wehrschuetz-Sigl E, Marold A, Wiesbauer H, Schoeftner R, Gewessler U, Kandelbauer A, Schiffer D, Schneider KP, Binder B, Schintler M, Guebitz GM. Analysis of myeloperoxidase activity in wound fluids as a marker of infection. Ann Clin Biochem. 2013 May;50(Pt 3):245-54. doi: 10.1258/acb.2011.010249. PMID 23404930
- [Background] Hasmann A, Gewessler U, Hulla E, Schneider KP, Binder B, Francesko A, Tzanov T, Schintler M, Van der Palen J, Guebitz GM, Wehrschuetz-Sigl E. Sensor materials for the detection of human neutrophil elastase and cathepsin G activity in wound fluid. Exp Dermatol. 2011 Jun;20(6):508-13. doi: 10.1111/j.1600-0625.2011.01256.x. Epub 2011 Apr 13. PMID 21488974
- [Background] Hasmann A, Wehrschuetz-Sigl E, Kanzler G, Gewessler U, Hulla E, Schneider KP, Binder B, Schintler M, Guebitz GM. Novel peptidoglycan-based diagnostic devices for detection of wound infection. Diagn Microbiol Infect Dis. 2011 Sep;71(1):12-23. doi: 10.1016/j.diagmicrobio.2010.09.009. Epub 2011 Mar 9. PMID 21388768
- [Background] Klebanoff SJ. Myeloperoxidase. Proc Assoc Am Physicians. 1999 Sep-Oct;111(5):383-9. doi: 10.1111/paa.1999.111.5.383. PMID 10519157
- [Background] Schiffer D, Blokhuis-Arkes M, van der Palen J, Sigl E, Heinzle A, Guebitz GM. Assessment of infection in chronic wounds based on the activities of elastase, lysozyme and myeloperoxidase. Br J Dermatol. 2015 Dec;173(6):1529-31. doi: 10.1111/bjd.13896. Epub 2015 Oct 29. No abstract available. PMID 25965963
- [Background] Heinzle A, Papen-Botterhuis NE, Schiffer D, Schneider KP, Binder B, Schintler M, Haaksman IK, Lenting HB, Gubitz GM, Sigl E. Novel protease-based diagnostic devices for detection of wound infection. Wound Repair Regen. 2013 May-Jun;21(3):482-9. doi: 10.1111/wrr.12040. Epub 2013 Apr 29. PMID 23627267
- [Background] Schiffer D, Tegl G, Heinzle A, Sigl E, Metcalf D, Bowler P, Burnet M, Guebitz GM. Enzyme-responsive polymers for microbial infection detection. Expert Rev Mol Diagn. 2015;15(9):1125-31. doi: 10.1586/14737159.2015.1061935. Epub 2015 Jul 16. PMID 26184576
- [Background] Tegl G, Schiffer D, Sigl E, Heinzle A, Guebitz GM. Biomarkers for infection: enzymes, microbes, and metabolites. Appl Microbiol Biotechnol. 2015 Jun;99(11):4595-614. doi: 10.1007/s00253-015-6637-7. Epub 2015 May 9. PMID 25952112